CLINICAL TRIAL: NCT03669289
Title: Enhanced Support for Behavioral Barriers to Learning: An Evaluation of the SCHOOL STARS (Supporting Child Health Outcomes, Optimizing Learning, Striving to Achieve Real Solutions) Program
Brief Title: Enhanced Support for Behavioral Barriers to Learning: An Evaluation of the SCHOOL STARS Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CIN001-SCHOOLSTARS
Record Dates: First submitted 2018-08-31; First posted 2018-09-13 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Disruptive Behavior Disorder, Childhood Onset; Attention Deficit Hyperactivity Disorder; Oppositional Defiant Disorder in Children; Disruptive Mood Dysregulation Disorder
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Pre-post within-subject design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enhanced model of primary care (Experimental)
  Interventions: Other: enhanced model of primary care

INTERVENTIONS:
Other: enhanced model of primary care — The SCHOOL STARS model of care includes pre-visit planning, standardized visit content, post-visit care coordination, and coordination between primary care and school.
  Other Names: SCHOOL STARS care model

SUMMARY:
This small pilot study will enroll children ages 5-12 years of age with disruptive behavior problems at school. These children and their families will be offered an enhanced model of primary care, which includes pre-visit record review, standardized content of primary care visits, post-visit care coordination by the primary care team, and coordination of services between the primary care team and the school. We hypothesize that children receiving this enhanced model of care will achieve better behavioral outcomes at both school and home.

ELIGIBILITY:
Inclusion Criteria:

* Student at a local public school
* Primary care patient at the Pediatric Primary Care Center (PPC) at CCHMC, or a CCHMC-affiliated school-based health center
* School disciplinary problems defined as: (1) any suspension from school within the last 2 school months and/or (2) frequent calls to the parent from school (1+ times per week x 1 month)
* Parent is in the contemplative, preparation, or action stage of readiness for starting medication or therapy if recommended by a healthcare provider for their child's behavior problems
* Student may or may not have an existing diagnosis of an externalizing behavioral health disorder, such as ADHD, Oppositional Defiant Disorder, or Disruptive Mood Dysregulation Disorder.

Exclusion Criteria:

* Non-English-speaking parent
* Enrolled in another ADHD study
* Severe developmental delay or autism
* Potential cardiac contraindications to starting stimulant medications without an EKG (personal or family history of heart disease in a child, family history of sudden death before age 50, family history of death due to heart disease before age 50, personal history of seizures, personal history of unexplained syncopal episodes)
* Patients who have an established relationship with a PPC Care Manager
* Patients who have seen the same primary care provider for the last two well child or behavior-related visits (unless approved/referred by that primary care provider)

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Child Behavior Checklist scores (externalizing subscale) | at enrollment and 3 months post-intervention
  parent-completed assessment of child behavior; T scores for the externalizing subscale range 0-100 with higher scores being worse

SECONDARY OUTCOMES:
Change in disciplinary referrals at school | 3 months pre-intervention to 3 months post-intervention
  number of times per week child was referred for disciplinary action at school
Change in calls to parent from school | 3 months pre-intervention to 3 months post-intervention
  number of calls per week to the parent from school about the child's behavior
Change in days of suspension from school | 3 months pre-intervention and 3 months post-intervention
  number of days child was suspended from school
Change in Vanderbilt Attention Deficit Hyperactivity Disorder Rating Scale scores | all historical data and all data up to 3 months post-intervention
  (for participants with ADHD); Total Symptoms Score for items 1-18 (inattentive and hyperactive symptoms); Range 0-54; Higher scores represent a worse outcome

OTHER OUTCOMES:
Referral adherence | from enrollment to 3 months post intervention
  percentage of referrals to behavioral therapy that result in a completed appointment

CONTACTS AND LOCATIONS:
Overall Officials: Courtney M Brown, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT03669289/ICF_000.pdf